CLINICAL TRIAL: NCT02435758
Title: Multicenter Study on Preservation Versus Excision of Denonvilliers Fascia in L-PANP Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Third Affiliated Hospital, Sun Yat-Sen University (Other)
Collaborators: Sixth Affiliated Hospital, Sun Yat-sen University (Other); Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Principal Investigator, Hongbo Wei, Assistant to the Dean, Third Affiliated Hospital, Sun Yat-Sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PED-PANP01
Record Dates: First submitted 2015-04-26; First posted 2015-05-06 (Estimated); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Rectal Cancer
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Preservation of Denonvilliers Fascia (Experimental): Preservation of Denonvilliers Fascia in Laparoscopy-assisted pelvic autonomic nerve preservation surgery with TME for male mid-low rectal cancer patients
  Interventions: Procedure: Preservation of Denonvilliers Fascia during L-PANP surgery
- Excision of Denonvilliers Fascia (No Intervention): Standard TME surgery (U-shaped excision of Denonvilliers fascia) in Laparoscopy-assisted pelvic autonomic nerve preservation surgery with TME for male mid-low rectal cancer patients

INTERVENTIONS:
Procedure: Preservation of Denonvilliers Fascia during L-PANP surgery — In this group, the patients accept L-PANP surgery, as well as preservation of Denonvilliers Fascia
  Arms: Preservation of Denonvilliers Fascia

SUMMARY:
TME (Total mesorectum excision) is the golden standard of radical resection for mid-low rectal cancer. However, the damage of pelvic autonomic nerve following with TME principle will lead to high incidence of urinary and sexual function disorder. PANP (pelvic autonomic nerve preservation) surgery played a role in decreasing incidence of urinary and sexual function disorder. However, 32%-44% patients still suffered from urinary and sexual function disorder when underwent open (O-PANP-TME) or laparoscopic PANP TME surgery (L-PANP-TME).

In the early stage of work, the investigators performed preservation of Denovilliers' fascia in L-PANP-TME to discuss the protection of urinary and sexual function of male mid-low rectal cancer patients. The results showed that preservation of Denovilliers' fascia in L-PANP-TME significantly decreased incidence of urinary and sexual function disorder. In order to further confirm the early work, the investigators design a multicenter randomized controlled clinical trial to compare differences in urinary and sexual function protection and long-term outcomes between preservation and excision of Denovilliers' fascia in L-PANP-TME.

ELIGIBILITY:
Inclusion Criteria:

1. Male, 20 < age (years) < 71, informed consent;
2. Pathological diagnosis of rectal adenocarcinoma;
3. Tumors from anal edge 6 ~ 12 cm (measured by rigid proctoscope);
4. Preoperative staging T1-4 (T1-2 for anterior rectal wall) N0-2M0 rectal cancer (AJCC- 7th);
5. R0 TME surgical results is expected;
6. Preoperative ECOG physical status score 0/1;
7. Preoperative ASA grade I ~ III;
8. Normal urinary function (Bladder residual urine<100ml), normal erection function (IIEF-5>21) and ejaculation function grading as I level.

Exclusion Criteria:

1. Complicated with acute ileus, perforation or hemorrhage;
2. Tumors with extensive invasion of surrounding tissues, TME not applicable; Imaging examination in regional integration intumescent lymph nodes (maximum diameter 3 cm or higher);
3. With other malignant diseases or with other malignant disease within 5 years; With other diseases need surgery;
4. A history of abdominal and pelvic major operation;
5. People with severe mental illness, or cannot be evaluated due to cultural or psychological factors;
6. No sexual life;
7. Critical organ dysfunction, unbearable surgery;
8. Unstable angina, myocardial infarction, cerebral infarction or hemorrhage within 6 months;
9. Systemic corticosteroids or immunosuppressive medication history within 1 month;
10. Pre-existent true incontinence or severe stress urinary incontinence.

Exit criteria:

1. Confirmed as M1 during or after operation;
2. Conversion to abdominoperineal resection (APR)
3. Postoperatively confirmed as invading rectal intrinsic fascia, or T3 for anterior rectal wall;
4. Intraoperative confirmed regional lymph node fusion conglobation cannot ensure R0 resection;
5. Infiltrating major blood vessel and unresectable;
6. Intraoperative finding other diseases need simultaneous surgery;
7. Preoperative emergent severe complications, cannot carry out the study treatment;
8. Emergency surgery is needed;
9. Into this study, at any stage of the initiative exit or discontinue treatment; Prove to implement the healer violates this research plan.

Ages: 20 Years to 71 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 262 (Actual)
Dates: Start 2015-04; Primary Completion 2020-05-06 (Actual); Study Completion 2023-06-15 (Actual)

PRIMARY OUTCOMES:
Urinary function | 14 days
  Urodynamic study and IPSS (International prostate symptom score) are used to assess urinary function
Sexual function | 14 days
  IIEF-5 (International questionnaire of erectile function-5) and Ejaculation function classification are used to assess sexual function

SECONDARY OUTCOMES:
Morbidity | 30 days
  incidence of postoperatvie complications
3-year overall survival rate | 36 months
  3-year overall survival rate
3-year recurrence pattern | 36 months
  3-year recurrence pattern
Mortality | 30 days
  incidence of postoperatvie deaths
5-year overall survival rate | 60 months
  5-year overall survival rate
5-year recurrence pattern | 60 months
  5-year recurrence pattern
3-year disease free survival rate | 36 months
  3-year disease free survival rate
5-year disease free survival rate | 60 months
  5-year disease free survival rate
Sexual function | 12 months
  International questionnaire of erectile function-5 (IIEF-5)
Sexual function | 12 months
  Ejaculation function classification
Urinary function | 12 months
  Urodynamic study and IPSS (International prostate symptom score) are used to assess urinary function

CONTACTS AND LOCATIONS:
Locations (1):
- The Third Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Wei B, Zheng Z, Fang J, Xiao J, Han F, Huang M, Xu Q, Wang X, Hong C, Wang G, Ju Y, Su G, Deng H, Zhang J, Li J, Chen T, Huang Y, Huang J, Liu J, Yang X, Wei H; Chinese Postoperative Urogenital Function (PUF) Research Collaboration Group. Effect of Denonvilliers' Fascia Preservation Versus Resection During Laparoscopic Total Mesorectal Excision on Postoperative Urogenital Function of Male Rectal Cancer Patients: Initial Results of Chinese PUF-01 Randomized Clinical Trial. Ann Surg. 2021 Dec 1;274(6):e473-e480. doi: 10.1097/SLA.0000000000004591. PMID 33234798